CLINICAL TRIAL: NCT01332773
Title: The ARTERY FIRST Approach for Resection of Pancreatic Head Cancer
Acronym: Artery first
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Jürgen Weitz, MD, MSc, Department of General, Visceral and Transplantation Surgery, University of Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNR-7
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2009-12

CONDITIONS: Pancreatic Head Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artery first group (Experimental): The basic principle of the "artery first" approach is the early identification of the SMA at its origin at the aorta with the further resection then being guided by its anatomic course.
  The dissection is carried cephalad along the aorta until the origin of the SMA is reached. The posterior and right aspect of the SMA is then dissected over a few centimeters. On the right side of the SMA a replaced or accessory right hepatic artery, if present, will be identified and preserved. This maneuver should be done, if infiltration of the SMA is suspected as the procedure can be terminated at this point. Once the situation at the SMA is assessed and resectability is confirmed resection will be done.
  Interventions: Procedure: Artery first procedure
- Conventional Group (Active Comparator): A wide Kocher manoeuver is performed to fully mobilize the duodenum and the head of the pancreas. The colonic mesentery on the right side is separated from the anterior surface of the duodenum and the head of the pancreas. The size of the tumor and its relation to the superior mesenteric artery, the celiac trunk, the mesentery, the portal vein, and the superior mesenteric vein is assessed. If resectability is given a Kausch-Whipple's resection is performed.
  Interventions: Procedure: No artery first procedure

INTERVENTIONS:
Procedure: Artery first procedure — early identification of SMA to evaluate infiltration
  Arms: Artery first group
Procedure: No artery first procedure — conventional exposure and preparation (Kocher's manoeuvre) before transection of pancreatic parenchyma
  Arms: Conventional Group

SUMMARY:
To show whether the artery first approach leads to equal or less rate of positive resection margins in pancreatic head cancer than the standard technique (ppWhipple only with standard Kocher's manoeuvre)

DETAILED DESCRIPTION:
This is a prospective non-randomized trial with two study groups. The trial is designed to show if the ARTERY FIRST approach reduces the rate of R1 resections in patients undergoing surgery for cancer of the pancreatic head.

After the diagnosis of cancer of the pancreatic head by clinical, laboratory and imaging evaluation patients who are scheduled for resection will be screened for inclusion into the trial. Informed consent is obtained at least on the day before surgery and patients meeting the eligibility criteria will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic head cancer (diagnosis by clinical, laboratory and radiological evaluation)
* Patients scheduled for curative resection
* No evidence of distant metastases
* Age equal or greater than 18 years
* Informed consent

Exclusion Criteria:

* Expected lack of compliance
* Impaired mental state or language problems
* patient having had neoadjuvant radiochemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Rate of R1 resections | up to 1.5 years
  positive resection margins as described by the pathologists of the University of Heidelberg

SECONDARY OUTCOMES:
Exploratory analyses | up to 1.5 years
  Exploratory analyses of frequencies of complications and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General, Visceral and Transplantation Surgery, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany